CLINICAL TRIAL: NCT03124771
Title: Accuracy of Noninvasive Hemoglobin Pulse Oximeter (Rainbow Resposable Adhesive Sensors)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TR23394-TP16171
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Results first posted 2017-06-06 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Rainbow Resposable Adhesive Sensors (Experimental): All subjects are enrolled into the test group and all subjects received the Rainbow Resposable Adhesive Sensors.
  Interventions: Device: Rainbow Resposable Adhesive Sensors

INTERVENTIONS:
Device: Rainbow Resposable Adhesive Sensors — Noninvasive Measurement of SpHb

SUMMARY:
In this study, the concentration of hemoglobin within the subject's blood will be reduced in a controlled manner by administering fluids intravenously. The accuracy of a noninvasive hemoglobin sensor(s) will be assessed by comparison to hemoglobin measurements from a laboratory analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18-40 years of age
* Weight of at least 110 lbs and less than 250 lbs or a BMI under 36 for subjects taller than 6 feet.
* Physical status of ASA I of II
* Able to read and communicate in English
* Has signed written informed consent
* Female, non pregnant. Female subjects will be provided with a pregnancy test free of charge.

Exclusion Criteria:

* Age less than 18 yrs and greater than 40 years
* Weight of less than 110 lbs or more than 250 lbs. or a BMI of 36 or greater for people over 6 feet tall.
* Hemoglobin less than 11 g/dL
* ASA physical status of III. IV, V.
* Pregnant
* Subject has known drug or alcohol abuse
* Subject has skin abnormalities affecting the digits such as psoriasis, eczema, angioma, scar tissue, burn, fungal infection, substantial skin breakdown, nail polish or acrylic nails.
* Subject has experienced a head injury with loss of consciousness within the last year.
* Subject has known neurological and psychiatric disorder that interferes with the subjects' level of consciousness.
* Known or concurrent chronic usage of psychoactive or anticonvulsive drugs within the last 90 days, or any use in the last 7 day (i.e. tricyclic antidepressants, MAO inhibitors, Lithum, neuroleptics, anxiolytics or antipsychotics, except SSRIs).
* Subject has any medical condition which in the judgment of the investigator, renders them inappropriate for participation in this study, such as Reynauds Syndrome.
* Systolic BP >140 mmHg or Diastolic BP > 100 mmHg.
* Baseline heart rate < 50 bpm.
* Inability to tolerate sitting still or minimal movement for up to 90 minutes
* Discretion of investigator

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2011-12-27 (Actual); Primary Completion 2012-04-03 (Actual); Study Completion 2012-04-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Rainbow Resposable Adhesive Sensor: All subjects are enrolled into the test group and all subjects received the Rainbow Resposable Adhesive Sensor.
Period: Overall Study
Arm/Group | Rainbow Resposable Adhesive Sensor
Started | 132
Completed | 132
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Rainbow Resposable Adhesive Sensors: All subjects are enrolled into the test group and all subjects received the Rainbow Resposable Adhesive Sensor.
Arm/Group | Rainbow Resposable Adhesive Sensors
Number analyzed (Participants) | 132
Age, Customized [Count of Participants; unit: Participants]
  18-40 years | 132
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 67

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Sensor by Arms Calculation
Description: Accuracy willl be determined by comparing the noninvasive hemoglobin measurement of the pulse oximeter to the hemoglobin value obtained from a blood sample and calculating the arithmetic root mean square(Arms) error value.
Time Frame: 1-5 hours
Measure: Number; unit: g/dL
Units Other Than Participants: data points
Arm/Group | Rainbow Resposable Adhesive Sensor
Number analyzed (Participants) | 132
Number analyzed (data points) | 1345
g/dL | 1.0

ADVERSE EVENTS:
Arm/Group | Rainbow Resposable Adhesive Sensor
Serious Adverse Events (participants affected / at risk) | 0/132
Other Adverse Events (participants affected / at risk) | 0/132

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes